CLINICAL TRIAL: NCT00688935
Title: Identification of Free-Running Rhythms in Blind Children
Brief Title: Young Blind Child Melatonin Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: eIRB 0714; n/a unfunded
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Blindness
Keywords: melatonin; circadian rhythms; sleep; sleep disorders
MeSH Terms: conditions — Blindness; Sleep Wake Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melatonin (Experimental): Subjects may opt to enroll in this treatment sub-study involving melatonin treatment (0.1 - 3 mg, daily) for up to 1 year, with a minimum of 6 weeks. Throughout treatment, subjects will continue their saliva, plasma, and/or urine sampling to test for treatment efficacy.
  Interventions: Biological: Melatonin

INTERVENTIONS:
Biological: Melatonin — 0.1-3 mg, daily, up to 1 year (minimum duration of 6 weeks)

SUMMARY:
The primary goal of this study is to identify the presence of desynchronized circadian rhythms in 25 children by measuring melatonin secretion in serial blood or saliva samples, and to rule out any primary sleep disorders.

DETAILED DESCRIPTION:
Subjects will complete 25-hours of hourly salivary, plasma sampling biweekly. Melatonin will be measured in urine, for children under the age of 3. Sleep and behavioral questionnaires will be completed by parents and/or teachers. This study involves an optional, 1-year melatonin treatment sub-study, in which the children will take 0.1 - 3mg daily. A second optional sub-study involves a study of the child's sleep through polysomnography, in order to identify possible sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-20 years
* Blindness for the past year (verified by an ophthalmologic exam), but otherwise in general good health.

Exclusion Criteria:

* Abnormal heart, lung, kidney, liver disease or a primary sleep disorder,
* Significant clinical abnormalities (other than blindness),
* Use of medications with known effects on melatonin metabolism (e.g. beta-adrenergic blocking drugs or tricyclic antidepressants).

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2005-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred J Lewy, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Sleep and Mood Disorders Lab, Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Palm L, Blennow G, Wetterberg L. Long-term melatonin treatment in blind children and young adults with circadian sleep-wake disturbances. Dev Med Child Neurol. 1997 May;39(5):319-25. doi: 10.1111/j.1469-8749.1997.tb07438.x. PMID 9236698
- [Background] Sack RL, Lewy AJ, Blood ML, Keith LD, Nakagawa H. Circadian rhythm abnormalities in totally blind people: incidence and clinical significance. J Clin Endocrinol Metab. 1992 Jul;75(1):127-34. doi: 10.1210/jcem.75.1.1619000.
- [Background] Tzischinsky O, Skene D, Epstein R, Lavie P. Circadian rhythms in 6-sulphatoxymelatonin and nocturnal sleep in blind children. Chronobiol Int. 1991;8(3):168-75. doi: 10.3109/07420529109063923. PMID 1794154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | Melatonin
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Melatonin
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Circadian Phase Marker, as Measured by the Melatonin Levels in Salivary, Plasma and/or Urine Serial Sampling.
Time Frame: every 2-4 weeks throughout the entire study
Population: as for baseline characteristics
Arm/Group | Melatonin
Number analyzed (Participants) | 0

2. Secondary Outcome: Polysomnography (Sleep Assessment)
Time Frame: 1 12-hour assessment any time during the study
Population: as for baseline characteristics
Arm/Group | Melatonin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Melatonin
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Analyses were not completed because, a unique provision in the American Recovery and Reinvestment Act (ARRA) of 2009 funding source unexpectedly prevented approval of a second year no-cost-extension in which completion of analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No